CLINICAL TRIAL: NCT05760820
Title: SES Children (SES Mini/SES Nxt) - A Digital Intervention for Children of Divorce
Acronym: SES Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Samarbejde efter Skilsmisse ApS (Unknown); The Agency of Family Law (Unknown); Aarhus Kommune (Other); Aabenraa Kommune (Unknown); Viborg Kommune (Unknown); Rudersdal Kommune (Unknown); Næstved Kommune (Unknown); Lyngby-Taarbæk Kommune (Unknown); Københavns Kommune (Other); Hvidovre Kommune (Unknown); Hillerød Kommune (Unknown); Herlev Kommune (Unknown); Gribskov Kommune (Unknown); Greve Kommune (Unknown); Glostrup Kommune (Unknown); Gladsaxe Kommune (Unknown); Furesø Kommune (Unknown); Favrskov Kommune (Unknown); Fredensborg Kommune (Unknown); Horsholm Municipality (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 504-0290/21-5000; 22-B-0105 (Other Grant/Funding Number: Helsefonden); 1045-00042B (Other Grant/Funding Number: Innovationsfonden); 514-0699/22-3000 (Other Grant/Funding Number: Data Protection Agency); 504-0290/21-5000 (Other: The Research Ethics Committee for Faculty of Science & Faculty of Health and Medical Sciences); 4956 (Other Grant/Funding Number: Egmont Foundation)
Record Dates: First submitted 2022-12-14; First posted 2023-03-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Parental Divorce; Parental Relationship Dissolution; Mental Health and Well-being
Keywords: Digital Intervention; Parental Divorce; Children age 3-17; Well-being; RCT Design; Quality of life
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention will be evaluated using a longitudinal ranodmized controlled trial study with a wait-list control design. Parents will be invited to the study and respond on behalf of children under the age of 11, while children aged 11 and older will respond to questions without parental assistance. Prior to baseline, parents (and all children of the parent) will be randomized (1:1) to either the intervention group (with access to the intervention) or the control group. Randomization will be blinded for participants only until the completion of the baseline questionnaire. All participants will be asked to complete questionnaires at 1- and 3-months post baseline. Those in the intervention group will gain immediate access to the digital intervention, while those in the control group will gain access after the 3-month follow-up questionnaire.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Access to the digital intervention post-baseline questionnaire and randomization.
  Interventions: Behavioral: SES Children (SES Mini & SES Nxt)
- Control Group (No Intervention): Control group will gain access to the digital intervention after the 3-month follow-up.

INTERVENTIONS:
Behavioral: SES Children (SES Mini & SES Nxt) — SES Children (SES Mini & SES Nxt) is a digital intervention aiming to develop children's self-efficacy and ability to overcome the challenges that come with a divorce and major life crises, thereby reducing the negative impacts of these on children's overall mental health and wellbeing. The intervention formatted to specific age groups between the ages of 3 and 17, and is relevant to all children whose parents have split up, regardless of whether they experience a higher or lower degree of conflict between the parents, a or higher or lower degree of strain from the judicial divorce.
  The intervention covers a variety of topics, including "when my parents fight", "a bonus family", "packing the overnight bag", "to live in two places", and "children's rights".
  Other Names: Samarbejde Efter Skilsmisse Children; Cooperation after Divorce Children
  Arms: Intervention Group

SUMMARY:
The overall aim of the SES Children (SES Mini/SES Nxt) - A Digital Intervention for Children of Divorce project is to develop the digital online intervention "SES Children (SES Mini & SES Nxt)", and test whether it reduces well-known negative consequences of divorce and major life crises among children and adolescents by employing a longitudinal RCT study design. SES Children (SES Mini & SES Nxt) is a digital intervention platform that seeks to develop the self-efficacy and ability of children to overcome the challenges that may come with a divorce and major life crises, thereby reducing the negative impacts of these on children's overall mental health and wellbeing. SES Children (SES Mini & SES Nxt) is a first of its kind and differs from existing interventions aimed at children in four crucial ways: 1) by being a comprehensive online intervention accessible via PC, smartphone, and tablet; 2) by being research-based and developed with the ambition of later scientific testing of its effect; 3) by offering early intervention to all children who experience parental divorce - not just children experiencing problems or conflicts in connection with parental divorce or who belong to certain age groups, and; 4) through its format and design, the intervention is adaptive to the individual child's needs and age and focuses on establishing real and lasting self-efficacy and behavioral change rather than only being informative and psycho-educational. Thus, unique to the solution are also unique methodological advances and knowledge related to digital interventions for children.

DETAILED DESCRIPTION:
The SES Children (SES Mini/SES Nxt) project consists of two main stages: 1) Development of the digital intervention, SES Children (SES Mini & SES Nxt), and 2) Testing the intervention.

Stage 1: The digital intervention has been developed. The content of the intervention is based on the research in child psychology and the factors suggested to be central to children's mental health and well-being (e.g., agency, prosociality, connection, normalization, and mentalization) as well as on the experiences and needs of professionals in the field. Specifically, collaboration with the Agency of Family Law was established, and the agency is considered the primary stakeholder in the field. The material was digitally implemented by experts in the field of digital learning.

Stage 2: The aim of the second stage is to assess the efficacy of the intervention in improving children´s study's primary and secondary outcomes. The intervention will be tested using a mixed-method design, including both a quantitative and a qualitative study methodology. This will take place in collaboration with the Agency of Family Law and Danish municipalities. Specifically, families will be invited to participate in the study by e-mail through the Agency of Family Law, Danish municipalities, and social media outreach. Individuals will receive an invitation letter, containing a short explanation of the study and a link to the study website, which contains a more thorough information sheet, eligibility questions, and an consent form.

The intervention will be evaluated using a two-armed, online, longitudinal randomized controlled trial (RCT), comparing an intervention group and a waitlist control group. Prior to baseline, participants will be randomized (1:1) to either the intervention group or the control group. Randomization will occur at the family-level, such that all members of the same family (the parent and the children that are signed up for study participation) will be in the same group. All participants will be asked to complete questionnaires at study inclusion (baseline), and at 1- and 3-months post baseline. Parents will be asked to respond to baseline questions covering basic socio-demographic variables and the outcome questionnaire. Parents will respond on behalf of children under the age of 11 (that is, we will obtain parent-report on children aged 3-10), while children aged 11 and older will respond to questions without parental assistance, as specified in the manual instructions for the outcome measures. Randomization will be blinded for the participant only until after the completion of the baseline questionnaire. After completion of the baseline questionnaires, those in the intervention group will gain immediate access to the digital intervention, while those in the control group will gain access after the 3-month follow-up questionnaire. The qualitative part of the evaluation will be conducted using semi-structured interviews with children and parents; these interviews will occur after the 1-month follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* be a custodial parent of at least one child between 3-17 year of age;
* be previously married and divorced or in a partnership and separated;
* have internet access;
* be able to write and read Danish.

Exclusion Criteria:

- not having a custodial child between 3-17 years of age.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Mental health and Well-being in Everyday Life - Emotional symptoms / problems | 3 months
  Strength and Difficulty Questionnaire (SDQ) The Strength and Difficulty Questionnaire (SDQ), emotional symptoms subscale, is the primary outcome. The subscale consists of 5 items that are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). The score is obtained by summing (appropriately reverse-scored) items together; scores can range from 0 to 10. Higher subscales scores indicate greater problems. The scale has been validated and normed to Danish children and adolescents aged 2-17 and has been used in numerous Danish and international studies (see also http://sdq.dk).
Mental health and Well-being in Everyday Life - Scale sum score | 3 months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents and has been found to be predictive of psychological and social functioning and (mal)adjustments in both the short term and in the longer run. The SDQ consists of 25 items that fall into five subscales: 1) Emotional symptoms, 2) Conduct problems, 3) Hyperactivity/inattention, 4) Peer relationships problem, and 5) Prosocial behavior. Items are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). A total difficulties score is generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0 to 40, with higher score, indicating more mental health and well-being related difficulties. The scale has been validated and normed to Danish children and adolescents aged 2-17 and has been used in numerous Danish and international studies.
Mental health and Well-being in Everyday Life - Impact score | 3-months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents. The SDQ contains an impact scale that assesses whether parents and children believe that the child has difficulties (in the areas of emotions, concentration, conduct, or social interactions), and if so, whether those difficulties interfere with the child's everyday life in terms of home life, friendships, classroom learning, and leisure activities. The impact supplement consists of 5 questions that are rated on a 4-point scale, with response options being "not at all" (0), "only a little" (0), "a medium amount" (1), and "a great deal" (2). The items are summed, and the resultant score can range from 0 to 10, with higher scores indicating greater impact of problems on daily life.

SECONDARY OUTCOMES:
Mental health and Well-being in Everyday Life - Conduct problems | 3 months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents and has been found to be predictive of psychological and social functioning and (mal)adjustments in both the short term and in the longer run. The conduct problems subscale consists of 5 items that are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). The score is obtained by summing (appropriately reverse-scored) items together; scores can range from 0 to 10. Higher subscales scores indicate greater problems.
Mental health and Well-being in Everyday Life - Hyperactivity/inattention | 3 months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents and has been found to be predictive of psychological and social functioning and (mal)adjustments in both the short term and in the longer run. The hyperactivity/inattention problems subscale consists of 5 items that are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). The score is obtained by summing (appropriately reverse-scored) items together; scores can range from 0 to 10. Higher subscales scores indicate greater problems.
Mental health and Well-being in Everyday Life - Peer relationships | 3 months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents and has been found to be predictive of psychological and social functioning and (mal)adjustments in both the short term and in the longer run. The peer relationship problems subscale consists of 5 items that are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). The score is obtained by summing (appropriately reverse-scored) items together; scores can range from 0 to 10. Higher subscales scores indicate greater problems.
Mental health and Well-being in Everyday Life - Prosocial Behavior | 3 months
  The Strength and Difficulty Questionnaire (SDQ) is used to assess mental health and well-being in everyday life among children and adolescents and has been found to be predictive of psychological and social functioning and (mal)adjustments in both the short term and in the longer run. The prosocial behavior subscale consists of 5 items that are rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). The score is obtained by summing (appropriately reverse-scored) items together; scores can range from 0 to 10. Higher scores indicate more positive social behavior.
Quality of Life - The QoL VAS | 3 months
  The Quality of My Life Questionnaire (QoML; Gong et al., 2007; Feldman et al., 2003 ) is used to assess quality of life (QoL) and health-related quality of life (HRQoL) as 2 separate constructs. For this study, the main outcome will be the QoL item, which is assessed using a visual analog scale. The QoL VAS asks "Overall, my life is . . ." Participants record their responses on a digital 100-mm VAS, which ranges from "the worst" (0) to "the best" (100); thus, the response range is from 0-100, with higher scores suggesting better QoL. The questions will only be completed by children age 11 to 17, at baseline, 1-month, and 3-month follow-up.
Somatization | 3 months
  Somatization is indicated by one question from the Strength and Difficulties Questionnaire, which assesses whether children experience headaches, stomach aches, or nausea (item 3 of the SDQ). The item is rated on a 3-point scale, with response options being "not true" (0), "somewhat true" (1), and "certainly true" (2). This item has previously been in a national cohort investigation of children's well-being in Denmark (Ottosen et al ., 2018).
Body size perception | 3 months
  We ask about perceptions of body size, with responses ranging from "much too thin" (1) to "much too fat" (5). This item was drawn from The Health Behaviour in School-aged Children (HBSC) study, which is a cross-national study of the health and health behaviors of adolescents across a large number of countries in Europe and North America, executed in collaboration with the World Health Organization (WHO) (Currie et al., 2104).
Sleep quality - difficulty falling asleep | 3-months
  Sleep quality is assessed by asking whether the child has had difficulties falling asleep during the last month. This item was also drawn from The Health Behaviour in School-aged Children (HBSC) study, which contained a section asking about health and well-being that included sleep (Currie et al., 2014, section 5.10; see also appendix 1, MQ55 of the HBSC study protocol). Participants are provided with the following response options: "never" (1), "a couple of times" (2), "almost every week" (3), "more than once a week" (4), and "almost every day" (5).

OTHER OUTCOMES:
Communicating needs | 3 months
  For the communicating needs domain, participants report about whether they have asked for help with money, new clothes, leisure activities, or other (instrumental support), whether they have communicated that they were upset (emotional support), or whether they have asked for advice or knowledge about something, if they needed it (informational support). Responses are provided on a 4-point rating scale; response options vary befitting with the question stem. For the first item, participants are provided with the following response options: "No and I haven't needed help" (0), "No, even though I have needed help" (1), "Yes, one time" (2), and "yes, multiple times" (3). Items are averaged to create a mean score that can range from 0 to 3; higher scores indicate greater frequency of communicating needs
Setting boundaries | 3 months
  For the setting boundaries domain, participants are asked whether they have spoken up and said no if parents have spoken badly about each other in front of the child, if the parents have had a verbal argument in front of the child, and if the parents have tried sending each other messages through the child. Responses are provided on a 4-point rating scale; response options vary befitting with the question stem. For the first item, participants are provided with the following response options: "No and they have not spoken badly about each other in front of me" (0), "No, even though they have not spoken badly about each other in front of me" (1), "Yes, one time" (2), and "yes, multiple times" (3). Items are averaged to create a mean score that can range from 0 to 3; higher scores indicate greater frequency of setting boundaries.
Connecting with an adult | 3 months
  With respect to the connecting with an adult domain, participants are asked how easy or difficult it has been for them to ask for help with money, new clothes, leisure activities, or other (instrumental support), whether they have communicated that they were upset (emotional support), or whether they have asked for advice or knowledge about something, if they needed it (informational support). Responses are provided on a 5-point rating scale, ranging from "very difficult" (1) to "very easy" (5). Items are averaged to create a mean score that can range from 1 to 5; higher scores indicate greater easy of connecting with an adult.
School attendance | 3 months
  School attendance will be measured with an items that examines whether and how many days the child has been absent from school or day care all day over the last 4 weeks (for baseline and the 1-month follow-up) or 8 weeks (for the 3-month follow-up). A percentage will be calculated for the full days of school attendance, with higher percentages indicate higher school attendance.
Parental Divorce Conflict | 3 months
  The DCS assesses parental conflict over three facets: (1) the domain dimension (areas of disagreements, e.g., child-rearing or finances), (2) the tactical dimension (the manner in which disagreements are resolved and managed), and (3) the attitudinal dimension (the general level of trust and hostility related to the former spouse). Participants respond to the items using a 4 to 6-point rating scale (response options vary by item stem). Items are summed together to create a score that can range from 0 to 27, such that higher scores indicate greater conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Martin Hald, PhD, Principal Investigator — University of Copenhagen; Camilla S Øverup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, København K, Denmark

IPD SHARING:
Plan to Share IPD: No